CLINICAL TRIAL: NCT07407296
Title: Multimodal Endoscopic Ultrasound in the Evaluation of the Nature of Indeterminate Upper Gastrointestinal Wall Thickening
Brief Title: Multimodal Endoscopic Ultrasound in the Evaluation of Indeterminate Upper Gastrointestinal Wall Thickening
Acronym: MM-EUS-UGIWT
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Taha Hussein Kawashty Abdelrahman, Assistent Lecturer at Tropical Medicine and Gastroenterology, Assiut University
Other Study IDs: MM-EUS-UGIWT
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Upper Gastrointestinal Wall Thickening
Keywords: Endoscopic Ultrasound in Upper Gastrointestinal Wall Thickening
MeSH Terms: interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Indeterminate Upper Gastrointestinal Wall Thickening
  Interventions: Procedure: Endoscopic ultrasound

INTERVENTIONS:
Procedure: Endoscopic ultrasound — Multimodal Endoscopic Ultrasound including; conventional B-mode EUS Assessment, doppler evaluation, EUS elastography and Selective EUS-Guided Fine-Needle Biopsy (EUS-FNB)

SUMMARY:
Multimodal endoscopic ultrasound can help to differentiate between benign (non-cancerous) and malignant (cancerous) causes of thickening of the upper digestive tract wall.

The main questions this study aims to answer are:

How accurate is multimodal endoscopic ultrasound in identifying the cause of upper digestive tract wall thickening?

Can using several ultrasound techniques together improve diagnosis when standard tests are unclear?

Participants are adults who have upper digestive tract wall thickening seen on scans such as computed tomography (CT) or magnetic resonance imaging (MRI).

Participants will:

Undergo upper endoscopy followed by endoscopic ultrasound and tissue sample taken during the procedure when needed followed by using biopsy results or clinical follow-up to confirm the final diagnosis

This study aims to improve early and accurate diagnosis and help guide proper treatment decisions for people with unexplained upper digestive tract wall thickening.

DETAILED DESCRIPTION:
Upper gastrointestinal wall thickening (UGIT) refers to the abnormal increase in the thickness of the gastrointestinal wall, which can be observed in various clinical conditions, including both benign and malignant diseases (1).

Abnormal gastric wall thickening can be caused by a wide range of benign and malignant conditions, and expedient diagnosis is required to commence the appropriate treatment (2, 3).

Traditional diagnostic approaches for evaluating UGIT rely primarily on cross-sectional imaging techniques such as contrast-enhanced computed tomography (CT) and magnetic resonance imaging (MRI). However, these modalities often lack sufficient spatial resolution to accurately characterize the individual layers of the gastrointestinal wall, particularly in cases of subtle mucosal or submucosal disease (4, 5).

Esophagogastroduodenoscopy (EGD) allows direct visualization of the mucosal surface and enables tissue sampling through conventional biopsies. Nevertheless, many pathological processes responsible for gastrointestinal wall thickening-such as gastric lymphoma, subepithelial tumors, linitis plastica, and infiltrative scirrhous carcinoma-originate in the deeper layers of the gastrointestinal wall (6).

EUS allows clear delineation of the gastrointestinal wall layers and surrounding structures. EUS-guided tissue acquisition using fine-needle biopsy (FNB) allows sampling of submucosal and muscular lesions that are inaccessible to conventional endoscopic biopsies (1).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with endoscopic or radiological (U/S, CT or MRI) evidence of upper GI wall thickening (esophagus, stomach, or duodenum) and defined based on established radiologic standards. A wall thickness by MSCT >5 mm in the oesophagus and stomach and >4 mm in the duodenum in accordance with accepted CT imaging criteria (4, 7).
* Written informed consent provided.

Exclusion Criteria:

* Patient refusal or inability to provide informed consent
* Uncorrectable coagulation disorder e.g prothrombin concentration <60%, INR >1.5 or platelet count <50,000/µL that cannot be corrected pre-procedure according to institutional guidelines.
* Presence of contraindications for endoscopy/sedation.
* Known diagnosis explaining wall thickening prior to EUS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with endoscopic or radiological (U/S, CT or MRI) evidence of upper GI wall thickening (esophagus, stomach, or duodenum) and defined based on established radiologic standards. A wall thickness by MSCT >5 mm in the oesophagus and stomach and >4 mm in the duodenum in accordance with accepted CT imaging criteria
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of multimodal EUS | one year

SECONDARY OUTCOMES:
EUS imaging patterns associated with various etiologies. | one year
Incremental diagnostic value of elastography. | one year
Diagnostic yield of EUS-guided tissue acquisition. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Taha Hussein El-sherif, Principal Investigator — Assit University
Locations (1):
- Assiut University, Asyut, Egypt, Egypt

REFERENCES:
- [Result] Desai R, Tagliabue J, Wegryn S, Einstein D. CT evaluation of wall thickening in the alimentary tract. Radiographics. 1991;11(5):771-83.
- [Result] Téllez-Ávila F, Duarte-Medrano G, Lopez-Arce G, Herrera-Mora D, Ramírez-Luna M, Valdovinos-Andraca F, et al. EUS-guided tissue samples for the diagnosis of patients with a thickened gastric wall and prior negative endoscopic biopsies. Acta Gastro-Enterologica Belgica. 2019;82.
- [Result] Macari M, Balthazar EJ. CT of bowel wall thickening: significance and pitfalls of interpretation. American Journal of Roentgenology. 2001;176(5):1105-16.
- [Result] Ergin M, Kıvrakoğlu F. Evaluation of Endoscopic Findings in Gastrointestinal Tract Wall Thickening Detected on kAbdominal Radiological Imaging: A Two-Center Retrospective Descriptive Study. Medicina. 2025;61(9):1699.
- [Result] Jung K, Park MI, Kim SE, Park SJ. Borrmann type 4 advanced gastric cancer: focus on the development of scirrhous gastric cancer. Clinical endoscopy. 2016;49(4):336-45.
- [Result] Chen T, Wu C, Lee C, Lai Y, Yang S. Endoscopic ultrasonography in the differential diagnosis of giant gastric folds. Journal of the Formosan Medical Association= Taiwan yi zhi. 1999;98(4):261-4.
- [Result] Giri S, Narayan J, Angadi S, Shah B, Ingle M, Tyagi U, et al. Role of endoscopic ultrasound-guided tissue acquisition for the diagnosis of gastric wall thickening: a retrospective study with meta-analysis. Annals of Gastroenterology. 2023;36(6):605.